CLINICAL TRIAL: NCT03850054
Title: AADI Glaucoma Shunt - a Quality Control Study
Status: Terminated | Type: Observational
Why Stopped: No further use of the divice at our department
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Anders H. Vestergaard, MD, PhD, Associate Professor, Odense University Hospital
Other Study IDs: 19/7009
Record Dates: First submitted 2019-02-04; First posted 2019-02-21 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Glaucoma
Keywords: AADI; glaucoma tube shunt
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: AADI glaucoma shunt — Implantation of the nonvalved AADI glaucoma shunt instead of the Bearveldt tube shunt, in eyes with intractable glaucoma.
  It is not a RCT study, but a prospective evaluation of the AADI device, and the study has been approved as a quality control study at the Department of Ophthalmology, at Odense University Hospital

SUMMARY:
To prospectively investigate the effect and safety of implantation of the AADI glaucoma tube in eyes with medically intractable glaucoma in the period 2019 to 2020, at the Department of Ophthalmology, Odense University Hospital.

The device will be implanted in eyes instead of the Bearveldt drainage device. Patients and data are prospectively registered to evaluate the effect and safety of the AADI device.

ELIGIBILITY:
Patients referred to glaucoma shunt implant (Baerveldt) will recieve the AADI glaucoma shunt

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Observational study, prospective, to evaluate the effect and safety of this new drainage device
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Change in IOP | Baseline and after 12 months
  Intraocular pressure before and after surgery
The change in number of IOP lowering drugs | Baseline and after 12 months
  Number of IOP lowering drugs before and after the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Dept. of Ophthalmology, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No
data will be deleted after use, as according to regulation

DOCUMENTS (1):
  • Study Protocol (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/54/NCT03850054/Prot_000.pdf